CLINICAL TRIAL: NCT07351409
Title: Immersive Virtual Reality as a Tool for Reducing Public Speaking Anxiety in Students Accessing the University Psychological Counseling Service: A Randomized Controlled Trial
Brief Title: VR-Counseling to Reduce Public Speaking Anxiety
Acronym: VR-Counseling
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calabria (Other)
Responsible Party: Principal Investigator, Francesco Craig, Associate professor, University of Calabria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RV-PSI_13/03/2023_n. 318
Record Dates: First submitted 2025-12-22; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: Anxiety and Distress; Anxiety; Anxiety Disease; Public Speaking Anxiety
Keywords: Public speaking anxiety; university counseling; Virtual Reality
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled, parallel-group interventional study with two independent arms (1:1 allocation): (1) an experimental group and (2) a control group. Both groups receive a brief standard counseling program consisting of six individual sessions delivered by trained clinicians within the University Psychological Counseling Service (UPCS). The experimental group receives the same counseling program plus two immersive VR modules delivered via 360° video scenarios: (a) VR-Exposure and Response Prevention (VR-ERP) for graded, controlled exposure to public-speaking situations, and (b) VR-Acceptance and Commitment Training (VR-ACT) providing ACT-consistent mindfulness and psychological flexibility exercises aimed at reducing arousal and enhancing coping. The control group receives counseling only (no VR).
  Outcomes are assessed at baseline (T0), post-treatment (T1), and follow-up (T2) to evaluate changes over time and between-group differences.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm: VR (360°) Modules (VR-ERP + VR-ACT) + Standard Counseling (Experimental): The experimental intervention includes two distinct VR-based training scenarios: (A) VR-ERP, designed to gradually expose students to anxiety-provoking situations to prevent avoidance responses, and (B) VR-ACT training, a consistent mindfulness training aimed at enhancing psychological flexibility and value-oriented behaviors. Participants in the experimental group, after VR-ACT training, go to standard counseling intervention.
  Interventions: Device: Exposure and Response Prevention (ERP); Device: Acceptance and Commitment Therapy (ACT) training
- Control Arm: Standard Counseling (No VR) (Active Comparator): Standard counseling sessions will be conducted by one psychotherapist for 6 consecutive weeks in 60-minute sessions.
  Interventions: Behavioral: Counseling program

INTERVENTIONS:
Device: Exposure and Response Prevention (ERP) — to simulate feared-anxiety-evoking scenarios, allowing both assessment and training for situationally induced anxiety to progressively promote desensitization to the anxiety-provoking stimuli
  Arms: Experimental Arm: VR (360°) Modules (VR-ERP + VR-ACT) + Standard Counseling
Device: Acceptance and Commitment Therapy (ACT) training — to provide an ACT-consistent mindfulness training targeting psychological flexibility processes, such as contact with the present moment, cognitive defusion, and acceptance, aimed at eliciting a grounding response within a digitally generated, safe environment.
  Arms: Experimental Arm: VR (360°) Modules (VR-ERP + VR-ACT) + Standard Counseling
Behavioral: Counseling program — Standard counseling sessions will be conducted by one psychotherapist for 6 consecutive weeks in 60-minute sessions.
  Arms: Control Arm: Standard Counseling (No VR)

SUMMARY:
Public Speaking Anxiety (PSA) is a common manifestation of social anxiety among university students that can negatively impact academic performance and psychological well-being. Virtual Reality (VR) based interventions combined with Cognitive Behavioral Therapy (CBT) represent a promising approach to address PSA by enabling controlled, gradual exposure to feared social situations through realistic simulations of audiences and settings. This randomized controlled trial will evaluate whether integrating VR sessions into standard psychological counseling provided by the University Psychological Counseling Service (UPCS) improves anxiety and PSA outcomes in university students compared with counseling alone.

Participants will be randomized to one of two groups: (1) a control group receiving standard psychological counseling intervention, or (2) an experimental group receiving psychological counseling supplemented with VR interventions delivered via immersive 360° video scenarios. The VR-based intervention includes a VR-Exposure and Response Prevention (ERP) module offering graded exposure to anxiety-provoking public speaking contexts, and a VR-Acceptance and Commitment Training (ACT) module aimed at enhancing mindfulness and psychological flexibility through guided experiential exercises. Psychological outcomes and physiological responses recorded during sessions will be analyzed to compare the effectiveness of VR-integrated counseling versus standard counseling alone. This study addresses the limited evidence on CBT combined with 360° video-based VR exposure for PSA in university students and introduces a novel VR-based ERP and ACT protocol tailored to a university counseling setting.

ELIGIBILITY:
Inclusion criteria are:

1. current enrollment at the university;
2. request for psychological counseling at the UPCS;
3. fluency in Italian;
4. provision of written informed consent;
5. the presence of at least moderate levels of anxiety and perceived stress, as indicated by scores on standardized assessment instruments. Specifically, scores between STAI scores from 35 to 50 and PRPSA scores from 85 to 110.

Exclusion criteria are:

1. current psychotic disorder;
2. acute suicidality;
3. severe substance dependence;
4. severe sensory or motor impairments that would prevent safe use of VR equipment;
5. inability to attend the planned sessions;
6. concurrent participation in other specialized psychotherapy programs.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-10-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Public Speaking Anxiety at VR Post-Treatment | Baseline (T0) and end of VR intervention sessions (T1, at the end of the 4-week intervention period).
  Change from baseline to post-treatment in public speaking anxiety as assessed by the Personal Report of Public Speaking Anxiety (PRPSA), comparing the experimental arm with the control arm.
  The PRPSA is a self-report questionnaire designed to measure anxiety specifically related to speaking in front of an audience. It assesses cognitive, physiological, and behavioral components of public speaking anxiety, capturing both anticipatory anxiety and anxiety experienced during performance. The scale consists of 34 items rated on a 5-point Likert scale, with response options ranging from 1 = strongly disagree to 5 = strongly agree. Items reflect feelings of tension and nervousness, physiological arousal, negative self-appraisal, and fear of audience evaluation. Total scores range from 34 to 170, with higher scores indicating greater levels of public speaking anx

SECONDARY OUTCOMES:
Heart Rate During Intervention Sessions | During VR intervention sessions, from session 1 (T0) through session 4 (T1 - end of the 4-week intervention period)
  Heart rate is continuously recorded during each intervention session to assess physiological arousal and recovery and to examine whether VR-supported counseling is associated with different within-session heart rate responses compared with counseling alone.
Heart Rate Variability During Intervention Sessions | During VR intervention sessions, from session 1 (T0) through session 4 (T1 - end of the 4-week intervention period)
  Heart rate variability is continuously recorded during each intervention session as an index of autonomic regulation and physiological recovery, and to compare within-session variability between VR-supported counseling and counseling alone.
Electrodermal Activity During Intervention Sessions | During VR intervention sessions, from session 1 (T0) through session 4 (T1 - end of the 4-week intervention period)
  Electrodermal activity is continuously recorded during each intervention session to assess sympathetic nervous system activation and physiological arousal during counseling, and to compare responses between treatment arms.
Skin Temperature During Intervention Sessions | During VR intervention sessions, from session 1 (T0) through session 4 (T1 - end of the 4-week intervention period)
  Skin temperature is continuously recorded during each intervention session as an indicator of peripheral physiological responses associated with stress and recovery, and to evaluate differences between VR-supported counseling and counseling alone.
Movement and Activity Levels During Intervention Sessions | During intervention sessions, from session 1 (T0) through session 4 (T1 - end of the 4-week intervention period)
  Movement and activity levels are continuously recorded during each intervention session to quantify physical activity and motion-related physiological responses and to compare within-session patterns between treatment arms.
Change From Baseline in Anxiety at VR Post-Treatment | During intervention sessions, from session 1 (T0) through session 4 (T1 - end of the 4-week intervention period)
  Change from baseline in anxiety assessed with the State-Trait Anxiety Inventory (STAI), Form Y, a widely used self-report questionnaire designed to measure two distinct dimensions of anxiety:
  (i) State Anxiety, a temporary emotional condition characterized by feelings of tension, apprehension, and heightened autonomic nervous system activity, reflecting how the respondent feels "right now, at this moment"; and (ii) Trait Anxiety, a relatively stable disposition to perceive situations as threatening and to respond with anxiety across time and contexts.
  Each subscale consists of 20 items rated on a 4-point Likert scale. Response options range from 1 = not at all to 4 = very much so for the State Anxiety subscale, and from 1 = almost never to 4 = almost always for the Trait Anxiety subscale. Total scores for each subscale range from 20 to 80, with higher scores indicating greater levels of anxiety.

OTHER OUTCOMES:
Change From Baseline in Public Speaking Anxiety at 3-Month Follow-Up | Baseline (T0) and 3-month follow-up (T2) (approximately 3 months after treatment completion).
  Change from baseline (T0) to the 3-month follow-up (T2) in public speaking anxiety (PSA). The experimental arm (VR intervention sessions) is expected to show greater sustained improvements at T2 compared with the control arm (brief standard counseling only).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calabria, Rende, CS, Italy

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data (IPD) underlying the results reported in publications will be made available upon reasonable request. Data will be shared in a de-identified format in accordance with applicable privacy regulations (e.g., GDPR).

REFERENCES:
- [Result] Reeves R, Curran D, Gleeson A, Hanna D. A Meta-Analysis of the Efficacy of Virtual Reality and In Vivo Exposure Therapy as Psychological Interventions for Public Speaking Anxiety. Behav Modif. 2022 Jul;46(4):937-965. doi: 10.1177/0145445521991102. Epub 2021 Feb 3. PMID 33533265
- [Result] Kampmann IL, Emmelkamp PM, Morina N. Meta-analysis of technology-assisted interventions for social anxiety disorder. J Anxiety Disord. 2016 Aug;42:71-84. doi: 10.1016/j.janxdis.2016.06.007. Epub 2016 Jun 18. PMID 27376634
- [Result] Kampmann IL, Emmelkamp PM, Hartanto D, Brinkman WP, Zijlstra BJ, Morina N. Exposure to virtual social interactions in the treatment of social anxiety disorder: A randomized controlled trial. Behav Res Ther. 2016 Feb;77:147-56. doi: 10.1016/j.brat.2015.12.016. Epub 2015 Dec 29. PMID 26752328
- [Result] Kahlon S, Lindner P, Nordgreen T. Virtual reality exposure therapy for adolescents with fear of public speaking: a non-randomized feasibility and pilot study. Child Adolesc Psychiatry Ment Health. 2019 Dec 27;13:47. doi: 10.1186/s13034-019-0307-y. eCollection 2019. PMID 31890004
- [Result] Huang J, Nigatu YT, Smail-Crevier R, Zhang X, Wang J. Interventions for common mental health problems among university and college students: A systematic review and meta-analysis of randomized controlled trials. J Psychiatr Res. 2018 Dec;107:1-10. doi: 10.1016/j.jpsychires.2018.09.018. Epub 2018 Sep 29. PMID 30300732
- [Result] Hendriks GJ, Janssen N, Robertson L, van Balkom AJ, van Zelst WH, Wolfe S, Oude Voshaar RC, Uphoff E. Cognitive behavioural therapy and third-wave approaches for anxiety and related disorders in older people. Cochrane Database Syst Rev. 2024 Jul 8;7(7):CD007674. doi: 10.1002/14651858.CD007674.pub3. PMID 38973756
- [Result] Donnelly MR, Reinberg R, Ito KL, Saldana D, Neureither M, Schmiesing A, Jahng E, Liew SL. Virtual Reality for the Treatment of Anxiety Disorders: A Scoping Review. Am J Occup Ther. 2021 Nov 1;75(6):7506205040. doi: 10.5014/ajot.2021.046169. PMID 34817595
- [Result] Craig F, Colella GM, Tenuta F, Mauti M, Gravina A, Calomino ML, Plastina R, Polito A, Costabile A. From psychological wellbeing to distress: the role of psychological counseling interventions in university students. Front Psychol. 2025 Aug 8;16:1602009. doi: 10.3389/fpsyg.2025.1602009. eCollection 2025. PMID 40861352
- [Result] Copeland WE, McGinnis E, Bai Y, Adams Z, Nardone H, Devadanam V, Rettew J, Hudziak JJ. Impact of COVID-19 Pandemic on College Student Mental Health and Wellness. J Am Acad Child Adolesc Psychiatry. 2021 Jan;60(1):134-141.e2. doi: 10.1016/j.jaac.2020.08.466. Epub 2020 Oct 19. PMID 33091568
- [Result] Cerolini S, Zagaria A, Franchini C, Maniaci VG, Fortunato A, Petrocchi C, Speranza AM, Lombardo C. Psychological Counseling among University Students Worldwide: A Systematic Review. Eur J Investig Health Psychol Educ. 2023 Sep 14;13(9):1831-1849. doi: 10.3390/ejihpe13090133. PMID 37754472
- [Result] Gallego A, McHugh L, Penttonen M, Lappalainen R. Measuring Public Speaking Anxiety: Self-report, behavioral, and physiological. Behav Modif. 2022 Jul;46(4):782-798. doi: 10.1177/0145445521994308. Epub 2021 Feb 16. PMID 33593107
- [Result] Auerbach RP, Mortier P, Bruffaerts R, Alonso J, Benjet C, Cuijpers P, Demyttenaere K, Ebert DD, Green JG, Hasking P, Murray E, Nock MK, Pinder-Amaker S, Sampson NA, Stein DJ, Vilagut G, Zaslavsky AM, Kessler RC; WHO WMH-ICS Collaborators. WHO World Mental Health Surveys International College Student Project: Prevalence and distribution of mental disorders. J Abnorm Psychol. 2018 Oct;127(7):623-638. doi: 10.1037/abn0000362. Epub 2018 Sep 13. PMID 30211576
- See also: Related Info — https://www.unical.it/didattica/orientamento/counselling/progetto-pro-bene-comune/